CLINICAL TRIAL: NCT06034067
Title: Osseodensification Versus Conventional Drilling for Implant Site Preparation: a Randomized Controlled Trial
Brief Title: Osseodensification Versus Conventional Drilling for Implant Site Preparation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Maanas Shah, Lecturer, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBRU IRB-2021-61
Record Dates: First submitted 2023-08-27; First posted 2023-09-13 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Dental Implant Failed; Jaw, Edentulous, Partially; Edentulous Alveolar Ridge; Osseointegration Failure of Dental Implant
Keywords: osseointegration; bone density; osteotomy; primary stability
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Intervention Model Description: * Prospective, in which participants will be recruited and then followed up throughout a specified period of time.
  * Randomized, parallel designed, concurrent controlled trial with participants randomly allocated to either control or test groups.
  * Double-blinded as both the participants and outcome accessors of radiographic outcomes will be blinded to the intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: - Double-blinded as both the participants and outcome accessors of radiographic outcomes will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osseodensification (test) group (Experimental): Implant site preparation will be completed using osseodensification technique where tapered multifluted burs (Densah Burs; Versah, MI, USA) will be used as per manufacturer's instructions.
  Interventions: Procedure: Osseodensification osteotomy preparation
- Standard (control) group (Active Comparator): Implant site preparation will be completed using conventional drilling protocol technique where standardized drills provided by Straumann (Straumann®, Institute Straumann AG, Basel, Switzerland)) will be used as per manufacturer's instructions.
  Interventions: Procedure: Standardized osteotomy preparation

INTERVENTIONS:
Procedure: Osseodensification osteotomy preparation — The implant site will be prepared by raising a mucoperiosteal flap. Implant osteotomy will be prepared by using osseodensification technique using Versah burs and a dental implant will be placed. The flaps will then be replaced and sutured with 4/0 polyglycolic acid interrupted and mattress sutures.
  Other Names: Densah® burs, Versah co., USA
  Arms: Osseodensification (test) group
Procedure: Standardized osteotomy preparation — The implant site will be prepared by raising a mucoperiosteal flap. Implant osteotomy will be prepared by using either conventional surgical drills provided by Straumann implant systems and a dental implant will be placed. The flaps will then be replaced and sutured with 4/0 polyglycolic acid interrupted and mattress sutures.
  Other Names: Straumann® Twist Drills, Straumann, Switzerland
  Arms: Standard (control) group

SUMMARY:
A total of 34 participants, who require replacement of an anterior or posterior single tooth with dental implant, will be randomly allocated to two equal sized groups. In the control group, the osteotomy site preparation will be prepared by using conventional surgical drills, while the test group site preparation will involve the use of Densah™ Burs (Versah Co., LLC., USA) as per the osseodensification protocol. In addition to evaluating implant stability, the trial will also report on implant and patient outcomes at various time points.

DETAILED DESCRIPTION:
Osseodensification technique has demonstrated increased primary stability and increased bone mineral density around the osteotomy site. The implants placed into osseous densification osteotomies have shown significant increase in insertion and removal torque values. This technique also burnishes bone along the inner layer of the osteotomy site and create a condensed layer of autografted bone along the periphery and apex of the implant. This would, in turn, increase the bone-implant contact enhancing the insertion torque values, and thus, primary implant stability. This new technique has not only shown increased primary implant stability when compared with conventional drilling, but also, shown to have similar clinical safety to conventional methods of osteotomy site preparation. Although osseodensification has been reported to enhance the clinical outcomes of implants by increasing primary stability, its long-term effects on implant stability measurements and implant survival rates are still not clear. The purpose of the present randomized controlled trial is to evaluate the stability of implants placed in sites prepared with either conventional drilling or osseodensification and report on implant and patient outcomes at various time points.

Objectives:

The aims of the randomized controlled trial are:

* To evaluate implant stability as measured by implant stability quotient (ISQ).
* To evaluate the clinical, radiographic outcomes and implant survival rates.
* To evaluate the need for additional bone augmentation at the time of implant placement.
* To evaluate changes in peri-implant marginal bone level.
* To evaluate bone quality as estimated by clinicians during osteotomy preparation.
* To evaluate biological and technical complications during the follow-up period.
* To evaluate patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over.
* Require replacement of an anterior or posterior single tooth with dental implant.
* Controlled oral hygiene (full-mouth plaque and bleeding scores ≤ 25% at baseline).
* Good compliance and commitment to attend follow-up review appointments.
* Willing to provide informed consent.

Exclusion Criteria:

* Localized / generalized periodontitis.
* Bone metabolic disease and/or taking medications that affect bone metabolism.
* Long term use of non-steroidal anti-inflammatory medications.
* History of malignancy, radiotherapy or chemotherapy.
* Pregnant or lactating women.
* Severe bruxism or parafunctional habits.
* Participants, who have controlled medical condition or smokers, will not be excluded in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Implant stability quotient (ISQ values) using resonance frequency analysis | Upto 36 months
  Resonance frequency analysis (RFA) will be used to determine stability (the level of osseointegration) in dental implants. The stability will be presented as an implant stability quotient (ISQ) value. The measurements will be recorded at time of implant placement, delivery of implant restoration (baseline), one year of implant restoration and annually up to three years using resonance frequency analysis.
Implant failure rate | Upto 36 months
  Implant failure rate will be assessed clinically after one year of implant restoration and annually up to three years.

SECONDARY OUTCOMES:
Changes in peri-implant marginal bone level (in mm) | Upto 36 months
  Changes in peri-implant marginal bone level will be assessed at implant placement, delivery of implant restoration (baseline), one year of implant restoration and annually up to three years using standardized peri-apical radiograph. The changes in peri-implant marginal bone levels will be recorded in millimeters
Descriptive evaluation of biological and technical complications associated with dental implant restorations | Upto 36 months
  Descriptive evaluation of biological and technical complications will be recorded during the follow-up period
Patient postoperative experience ( visual analogue scale ) | Upto 10 days
  Patient postoperative experience will be assessed using visual analogue scale during the first week following implant placement; the scale consists of a 10cm line, with end points representing 0 ('no pain') and 10 ('unbearable/worst pain'). The participant will be asked to place a mark on he line indicating the level of pain that he/she experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Maanas S Shah, BDS MSD CAGS, Principal Investigator — Mohammed Bin Rashid University of Medicine and Health Sciences
Locations (1):
- Dubai Dental Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albrektsson T, Zarb GA. Current interpretations of the osseointegrated response: clinical significance. Int J Prosthodont. 1993 Mar-Apr;6(2):95-105. PMID 8329101
- [Background] Atieh MA, Alsabeeha NH, Faggion CM Jr, Duncan WJ. The frequency of peri-implant diseases: a systematic review and meta-analysis. J Periodontol. 2013 Nov;84(11):1586-98. doi: 10.1902/jop.2012.120592. Epub 2012 Dec 13. PMID 23237585
- [Background] Atsumi M, Park SH, Wang HL. Methods used to assess implant stability: current status. Int J Oral Maxillofac Implants. 2007 Sep-Oct;22(5):743-54. PMID 17974108
- [Background] Buser D, Halbritter S, Hart C, Bornstein MM, Grutter L, Chappuis V, Belser UC. Early implant placement with simultaneous guided bone regeneration following single-tooth extraction in the esthetic zone: 12-month results of a prospective study with 20 consecutive patients. J Periodontol. 2009 Jan;80(1):152-62. doi: 10.1902/jop.2009.080360. PMID 19228101
- [Background] Buser D, von Arx T, ten Bruggenkate C, Weingart D. Basic surgical principles with ITI implants. Clin Oral Implants Res. 2000;11 Suppl 1:59-68. doi: 10.1034/j.1600-0501.2000.011s1059.x. PMID 11168257
- [Background] Di Stefano DA, Perrotti V, Greco GB, Cappucci C, Arosio P, Piattelli A, Iezzi G. The effect of undersizing and tapping on bone to implant contact and implant primary stability: A histomorphometric study on bovine ribs. J Adv Prosthodont. 2018 Jun;10(3):227-235. doi: 10.4047/jap.2018.10.3.227. Epub 2018 Jun 12. PMID 29930793
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Huwais S, Meyer EG. A Novel Osseous Densification Approach in Implant Osteotomy Preparation to Increase Biomechanical Primary Stability, Bone Mineral Density, and Bone-to-Implant Contact. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):27-36. doi: 10.11607/jomi.4817. Epub 2016 Oct 14. PMID 27741329
- [Background] Inchingolo AD, Inchingolo AM, Bordea IR, Xhajanka E, Romeo DM, Romeo M, Zappone CMF, Malcangi G, Scarano A, Lorusso F, Isacco CG, Marinelli G, Contaldo M, Ballini A, Inchingolo F, Dipalma G. The Effectiveness of Osseodensification Drilling Protocol for Implant Site Osteotomy: A Systematic Review of the Literature and Meta-Analysis. Materials (Basel). 2021 Feb 28;14(5):1147. doi: 10.3390/ma14051147. PMID 33671038
- [Background] Javed F, Ahmed HB, Crespi R, Romanos GE. Role of primary stability for successful osseointegration of dental implants: Factors of influence and evaluation. Interv Med Appl Sci. 2013 Dec;5(4):162-7. doi: 10.1556/IMAS.5.2013.4.3. Epub 2013 Dec 20. PMID 24381734
- [Background] Lioubavina-Hack N, Lang NP, Karring T. Significance of primary stability for osseointegration of dental implants. Clin Oral Implants Res. 2006 Jun;17(3):244-50. doi: 10.1111/j.1600-0501.2005.01201.x. PMID 16672018
- [Background] Meredith N. Assessment of implant stability as a prognostic determinant. Int J Prosthodont. 1998 Sep-Oct;11(5):491-501. PMID 9922740
- [Background] Sennerby L, Meredith N. Resonance frequency analysis: measuring implant stability and osseointegration. Compend Contin Educ Dent. 1998 May;19(5):493-8, 500, 502; quiz 504. PMID 9693511
- [Background] Sennerby L, Meredith N. Implant stability measurements using resonance frequency analysis: biological and biomechanical aspects and clinical implications. Periodontol 2000. 2008;47:51-66. doi: 10.1111/j.1600-0757.2008.00267.x. No abstract available. PMID 18412573
- [Background] Trisi P, Berardini M, Falco A, Podaliri Vulpiani M. New Osseodensification Implant Site Preparation Method to Increase Bone Density in Low-Density Bone: In Vivo Evaluation in Sheep. Implant Dent. 2016 Feb;25(1):24-31. doi: 10.1097/ID.0000000000000358. PMID 26584202
- [Background] Trisi P, Perfetti G, Baldoni E, Berardi D, Colagiovanni M, Scogna G. Implant micromotion is related to peak insertion torque and bone density. Clin Oral Implants Res. 2009 May;20(5):467-71. doi: 10.1111/j.1600-0501.2008.01679.x. PMID 19522976